CLINICAL TRIAL: NCT01872923
Title: Dose Escalating Study to Evaluate the Tolerability, Efficacy and Safety of Amphinex 0.125 mg/kg or Lower in Amphinex-based PCI of Bleomycin in Patients With Local Recurrence or Advanced/Metastatic, Cutaneous or Sub-cutaneous Malignancies.
Brief Title: Dose Escalating Study for Amphinex-based PCI of Bleomycin.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PCI Biotech AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCI 101/06 Extension; 2011-003750-80 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-06-07 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Cutaneous or Sub-cutaneous Malignancies
Keywords: Amphinex; PCI; Bleomycin; Cutaneous malignancies; Sub-cutaneous malignancies; Safety; Phase I; Photochemical Internalisation; Squamous Cell Carcinoma; Head and Neck cancer; Breast Cancer; HNSCC; SCCHN; Advanced or metastatic cancer; Dose finding
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis | interventions — Bleomycin; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amphinex based PCI of bleomycin (Experimental): The photosensitiser Amphinex is activated by Laser to enhance the effect of Bleomycin
  Interventions: Drug: Amphinex; Drug: Bleomycin; Device: Laser

INTERVENTIONS:
Drug: Amphinex — Photosensitiser
Drug: Bleomycin — Anticancer agent
Device: Laser — Laser that emits red light at 652 nm.
  Other Names: Ceralas PDT 652+/-3nm 2W" by CeramOptec GmbH CE0297

SUMMARY:
The primary goal of this extension study is to further investigate the tolerability and efficacy in a phase I setting in order to see whether lower doses than the initial study dose of 0.25 mg/kg bw Amphinex in Amphinex-based PCI of bleomycin will show a comparable or improved safety and tolerability profile in combination with comparable signs of efficacy.

DETAILED DESCRIPTION:
Use of Amphinex for the enhancement of Bleomycin at the intracellular target. The photosensitizer Amphinex is activated by Laser Light at 652 nm.

Superficial lesions (cutaneous or subcutaneous) was treated with the laser light after administration of Amphinex and Bleomycin according to time scheduled provided.

Safety and preliminary effect data where evaluated at a lower dose than explored in the preceeding dose escalating study with Amphinex.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female aged 18 years or above who have given written informed consent

  * Skin type I- IV according to the Fitzpatrick skin classification (see Appendix G)
  * With a diagnosis of local recurrence or advanced/metastatic, cutaneous or subcutaneous malignancy
  * Lesion measurement must not be done more than 2 weeks before the beginning of treatment. More than one field with lesion can be illuminated, but care must be taken to avoid overlap of the fields illuminated
  * Have discontinued any other investigational therapy or radiotherapy for at least 2 weeks prior to administration of Amphinex at the baseline visit, and have recovered from the acute effects of therapy
  * Have discontinued cytostatic or cytotoxic therapies with at least 6 half life cycles of the agent prior to administration of Amphinex at the baseline visit
  * Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Scale (see Appendix D)
  * Clinically assessed as eligible for bleomycin chemotherapy
  * Have a predicted life expectancy of at least 3 months
  * Geographic proximity that allow adequate follow-up
  * If female: have had childbearing potential either terminated by surgery, radiation, or menopause or attenuated by the use of an approved contraceptive method during and for 3 months after the trial
  * If male: have had reproductive potential either terminated or attenuated by the use of an approved contraceptive method during and for 3 months after the trial.

Exclusion Criteria:

* Have received prior PCI

  * Tumours known to be eroding into a major blood vessel in or adjacent to the illumination site
  * Planned surgery in first 28 days after treatment, except for planned surgical removal of the treated lesion
  * Planned dentist appointments in first 28 days after treatment
  * Anticancer therapy within the first 28 days after treatment
  * Therapy with drugs that induce light sensitivity (e.g. tetracyclines, sulfonamides, phenothiazines, sulfonylurea, hypoglycemic agents, thiazide diuretics, and griseofulvin) within the first 14 days after treatment
  * Co-existing ophthalmic disease likely to require slit-lamp examination within the first 28 days after treatment
  * History of hypersensitivity/anaphylactic reactions
  * Previous cumulative dose of Bleomycin received over 200 000 IE
  * Known allergy or sensitivity to photosensitisers
  * Known allergy to Cremophor
  * Known allergy to bleomycin
  * Conditions contraindicated for bleomycin treatment (lung infection, impaired pulmonary function)
  * Conditions that worsen when exposed to light (including porphyria)
  * Conditions associated with a risk of poor protocol compliance
  * Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To assess the combined tolerability and efficacy of Amphinex 0.125 mg/kg or lower in Amphinex-based PCI of bleomycin | From Baseline to 3 months
  Maximal pain during the procedure will be recorded immediately after the procedure on a 10 centimetre visual analogue scale (VAS). Pain will also be recorded 24 hours after the illumination and on day 4. The end-points of the VAS will be "no pain" and "unbearable pain
  A formal efficacy analysis is not appropriate for this trial. The response data will be documented by descriptive summary tables. No statistical comparison of dose levels will be done. Fluorescence measurements over time and lesion response evaluation according to RECIST (see Appendix E) will be presented for APT and PP stratified by dose level.

SECONDARY OUTCOMES:
To evaluate the safety of Amphinex 0.125 mg/kg or lower in Amphinex-based PCI of bleomycin. | From Baseline to 3 months
  * Summaries of the adverse event rates and laboratory changes from baseline stratified by dose level.
  * Listings and frequency tables categorizing laboratory and non-laboratory adverse events by maximum CTCAE toxicity grade and relationship to study drug.
  * Pain measurement, fluorescence measurement, skin photosensitivity measurement

OTHER OUTCOMES:
To determine the pharmacokinetics of Amphinex 0.125 mg/kg or lower in Amphinex-based PCI of bleomycin. | From Baseline to 3 months
  Plasma samples for pharmacokinetic (PK) evaluation will be collected from patients and the presence of Amphinex and/or other unidentified metabolites will be assessed using a validated analytical method
  Systematic skin photosensitivity tests will be carried out using a white light source with an emission spectrum that, relatively to the luminance and within +/- 50%, excites Amphinex with the same efficiency as sunlight. The luminance will be 500 lux, which is comparable to bright indoor light, and 100.000 lux, which is comparable to direct sunlight. The phototoxic reaction will be scored at specific time points following the light exposure (see the study flowchart Appendix B). This information will be used to predict the degree of photosensitivity of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, MD, Principal Investigator — UCLH
Locations (1):
- University College London Hospital, London, United Kingdom